CLINICAL TRIAL: NCT00195325
Title: A Phase 1 Dose Escalation Study of TTI-237 Administered Intravenously (IV) Once Weekly in Subjects With Advanced Malignant Solid Tumors.
Brief Title: Study Evaluating TTI-237 in Advanced Malignant Solid Tumors.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 3162K1-100
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-03-26 (Estimated); Status verified 2007-03

CONDITIONS: Tumors; Neoplasms
Keywords: Advanced Malignant Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — cevipabulin

INTERVENTIONS:
Drug: TTI-237

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and MTD (maximum tolerated dose) of TTI-237 for the treatment of subjects with advanced malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of malignant solid tumor with measurable disease
* Life expectancy of at least 12 weeks
* ECOG (The Eastern Cooperative Oncology Group scale) performance status of 0, 1, or 2

Exclusion Criteria:

* Recent major surgery, radiation therapy or anti-cancer treatment
* History of any other prior malignancy within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2005-08

PRIMARY OUTCOMES:
To determine safety, tolerability, and MTD of TTI-237 - patients are monitored during the duration of their participation on the trial.

SECONDARY OUTCOMES:
Preliminary pharmacokinetics (during cycle 1) and anti-tumor activity of TTI-237 (approximately every 8 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (3):
- United States (3):
  - Lexington, Kentucky
  - Cleveland, Ohio
  - Nashville, Tennessee